CLINICAL TRIAL: NCT04888364
Title: Cohort of the French Clinical Research Network for Parkinson's Disease (NS-PARK Cohort)
Brief Title: French Parkinson's Disease Cohort - NS-PARK
Acronym: NS-PARK
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-56; 2019-A01929-48 (Registry Identifier: RCB ID)
Record Dates: First submitted 2021-04-19; First posted 2021-05-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Genetics
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Biosampling is optional and includes:
  * biosamples specifically collected for this research: blood samples (for DNA extraction and storage, peripheral white blood cells, and plasma); skin biopsy for isolation, culture and storage of fibroblasts; urine; saliva;
  * biosamples collected in clinical routine, part of it being stored for research purposes: CSF, salivari accessory gland biopsies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of NS-PARK cohort are to describe the natural history of Parkinson's disease (PD), and to propose patients stratification models based on PD pathophysiological mechanisms. Patients are included at all PD expert centers in France. Standardized demographic, diagnosis, motor and non-motor symptoms evaluation, and treatment information are collected, and clinical data are updated at each visit of the patient at the center. A blood sampling is perform at baseline for genetic testing and implement an associated biocollection.

DETAILED DESCRIPTION:
The national clinical research network for Parkinson's disease (NS-PARK/FCRIN) reassembles all expert centers in Parkinson's disease (PD) in France. Its aim is to promote clinical research in Parkinson's disease and movement disorder, to better understand the pathophysiology of PD, foster the development of new therapeutic strategies, and move towards personalized medicine. To help centers for prescreening, a national registry of PD patients followed in each centers has been implemented in 2016 to collect minimal relevant clinical information of patients followed in each center including demographic data, age at diagnosis, standardized motor and non-motor symptoms evaluation, and treatment. Data are updated at each visit of the patient in the center. De facto, this registry became a longitudinal cohort of PD patients followed in NS-PARK centers. In 2020, NS-PARK received funding to associate a biocollection to this clinical cohort.

The aim of NS-PARK cohort are to describe the natural history of PD progression in clinical routine in France, to develop new models of PD describing the different progression profiles, and to propose patients stratification based on PD pathophysiological mechanisms. The cohort will also serve as a platform to discover new PD genes and genetic modifiers of disease progression or response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to UK PD brain bak criteria
* OR diagnosis of parkinsonian syndrome: multiple system atrophy, progressive supranuclear palsy, dementia with Lewy body, or corticobasal syndrom
* OR Subjects at risk of PD defined as :

No symptom or diagnosis of Parkinson's disease nor parkinsonian syndrome, and relative to a patient with a diagosis of PD or parkinsonian syndrome, or carrier of a known mutation responsible for a genetic form of PD or patient with a diagnosis of idiopathic REEM sleep disorder or prodromal form of PD as defined by MDS criteria (Berg et al., 2015)

AND for all participants

* Affiliated to social security
* Age > 10 years

Exclusion Criteria:

* Subject under legal protection
* Subject who do not consent to the research
* for the optional skin biopsy only: clinically significant coagulation abnormalities or anticoagulant treatment

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients followed at one expert center for PD or associated centers in France.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease progression | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Hoehn and Yahr score change
Motor and non-motor complications | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Occurence of motor (dyskinesia or motor fluctuations) or non-motor (dementia, dysautonomia, behavioral or psychiatric disorders, sleep disorders, falls, ...) complication
Modification of antiparkinsonian treatment doses | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Modification of antiparkinsonian treatment during follow-up will be measured as levodopa equivalent daily doses

SECONDARY OUTCOMES:
Predictive factorsof PD progression: motor or non motor symptoms | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Motor or non motor symptoms as measured by MDS-UPDRS scores will be used as predictive factors for primary outcomes
Predictive factors of PD progression: genetic variants | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Genetic variants in PD genes or the Genetic PD risk score will be used as predictive factors for primary outcomes.
Predictive factors of PD progression: brain imaging markers | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Brain imaging makers (iron or neuromelanine content of the substantia nigra) will be used as predictive factors for primary outcomes
Clusters of patients with similar disease progression profiles | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Clustering analyses will be performed on disease progression markers (Hoehn and Yahr score, MDS-UPDRS scores, and doses of treatment (levodopa equivalent daily doses)) to identify homogeneous groups of patients (clusters) sharing similar disease progression profiles.
Clusters of patients with similar genetic and disease progression profiles | through the end of follow-up in the cohort, at least 2 years, and average of 5 years
  Co-clustering analysis of disease progression markers (Hoehn and Yahr score, MDS-UPDRS scores, and doses of treatment (levodopa equivalent daily doses)) and genetic markers (variants in PD genes or the Genetic PD risk score).
Genetic mutations associated with familal forms of PD | through study completion, 15 years
  Genetic mutations will be screened by different methods (gene panels, whole exome or whole genome) in familial forms of PD. Mutations co-segregated with PD will be considered as potentially associated with the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe MD CORVOL, PU-PH, Principal Investigator — UMRS 1127
Locations (1):
- Centre 01 Paris, Paris, France

REFERENCES:
- [Derived] Lanore A, Januel E, Bertille N, Fabbri M, Mariani LL, Mangone G, Sambin S, Menon PJ, Tir M, Bereau M, Meissner WG, Thiriez C, Marques A, Remy P, Dupont G, Moro E, Defebvre L, Houeto JL, Thobois S, Azulay JP, Geny C, Frismand S, Damier P, Giordana C, Castelnovo G, Ansquer S, De Maindreville AD, Drapier S, Maltete D, Tranchant C, Rascol O, Tubach F, De Rycke Y, Corvol JC; French NS-Park Network. Motor and Non-motor Complications Following Different Early Therapies in Parkinson's Disease: Longitudinal Analysis of Real-Life Clinical and Therapeutic Data from the French NS-PARK Cohort. CNS Drugs. 2025 Sep;39(9):879-891. doi: 10.1007/s40263-025-01193-5. Epub 2025 May 25. PMID 40415148